CLINICAL TRIAL: NCT02714257
Title: Integrating Patient-Centered Exercise Coaching Into Primary Care to Reduce Fragility Fracture
Brief Title: Working to Increase Stability Through Exercise
Acronym: WISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); University of Pittsburgh (Other); Temple University (Other); Johns Hopkins University (Other); Columbia University (Other); University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Christopher Sciamanna, MD, MPH, Prof. Medicine and Public Health Sciences, Division Chief Population Health Research and Development, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-3576; PCS-1406-18325-EXT (Other: PCORI)
Record Dates: First submitted 2016-02-22; First posted 2016-03-21 (Estimated); Results first posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Fractures, Bone
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced Usual Care - control group (No Intervention): Participants will receive enhanced usual care by reviewing three printed pamphlets on fall risks and recommendation to exercise. In addition, to maximize patient safety, the investigators will communicate the baseline bone density results (measured by Dual-energy X-ray absorptiometry, DXA) to the patient's primary care provider, and any critical values of a baseline measure.
- Enhanced Usual Care plus Exercise Coaching Intervention (Experimental): Participants will receive the three printed pamphlets on fall risks and exercising in groups (same as the controls) plus: (1) an exercise program that includes strength, balance, and aerobic exercises; (2) an exercise coach that provides in-person and telephone support/feedbacks to enhance participation in the exercise program; and (3) regular progress reports sent by coaches by fax/Electronic Health Records every 4 months, to communicate the patient's progress.
  Interventions: Behavioral: Enhanced Usual Care plus Exercise Coaching

INTERVENTIONS:
Behavioral: Enhanced Usual Care plus Exercise Coaching — For month one of the exercise intervention the investigators will conduct only strength and a few balance exercises to rehabilitate the participants. After the first month, and once the participants feel comfortable, the investigators will incorporate aerobic and additional balance exercises. The investigators will personalize participant programs based on baseline levels and increase them gradually. The exercise session will be conducted 50 minutes 3 times a week. Between sets there is a 60-second break.
  Every month the coach will record steps from the pedometer and record patient adherence to exercise sessions, and every 2 months the coach will measure strength and will track resistance band color from the exercise trackers.
  For the individuals exercising at home, the investigators will distribute the exercise Digital Versatile Disc (DVDs) every 9 months and the coach will continue to contact them, just as if they were joining the group. Coaches will encourage group participation.
  Arms: Enhanced Usual Care plus Exercise Coaching Intervention

SUMMARY:
The investigators propose a 36-month multi-center randomized effectiveness trial to compare the impact of an Enhanced Usual Care (Control) intervention, with Exercise Coaching (Exercise), on Fragility Fractures and Serious Fall-Related Injuries (FF/SFRI) in patients with a previous fragility fracture (FF).

The investigators will also examine the impact of the intervention on several secondary outcomes like: loneliness, physical function, and bone strength. The investigators will do this by following a Pragmatic trial design: 1) limiting exclusions to increase representativeness, 2) limiting research contacts (average 30 min/year) and 3) limiting measures to those practicable for use in usual care.

DETAILED DESCRIPTION:
The intervention will be held in churches, community centers, and senior residential facilities. Investigators will work with the exercise sites to recruit up to 125 individuals (5 per exercise site location) to serve as the Group leaders at each site location. Group leaders will be trained on the exercises and leadership roles to help lead the group. The investigators will ask them to come at least once per week, so the time commitment is minimal.

The investigators will be recruiting 1130 patients who have suffered a fragility fracture and will randomly assign them to one of two conditions: (A) Control Group - Enhanced Usual Care and (B) Intervention Group - Enhanced usual care plus Exercise coaching that includes in-person and phone coach contacts to encourage and support strength, balance and walking activities.

*Due to the COVID-19 pandemic, the in-person intervention was stopped in March of 2020 and a Zoom-based virtual intervention was introduced in April of 2020. Participants that join the zoom-based virtual intervention are lead by staffed exercise coaches.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 65 years old
* Previous Fragility Fracture (FF) in past 10 years.
* Able to speak and understand English.
* Participants will need to be willing to try exercising and agree to annual follow-up measurements.

Exclusion Criteria:

If the answer to the following questions are "yes", the investigators will exclude the participant from the study Do you feel pain in your chest, neck, jaw, or arms at rest, during your daily activities of living, OR when you do physical activity? Have you ever been told by a health professional that you should not exercise OR exercise only when supervised by a professional?

If the answer to the following questions are "yes", the investigators will contact physician for permission Do you experience unpleasant awareness of a forceful or rapid heart rate? Do you experience unreasonable breathlessness? Do you experience dizziness fainting or blackouts? Do you experience ankle swelling? Do you have burning or cramping sensation on your lower legs when walking short distances? Do you have diabetes?

Has a doctor, nurse or health professional ever told you that you had any of the following? Weak or failing kidneys? A heart attack, also called a myocardial infarction? Angina or coronary heart disease? A stroke? Any kind of heart condition or heart disease other than the ones I just asked about?

Unable to obtain primary care provider consent (if required based on questions above)

If the participant answer "NO" to the following question: Is it ok if the investigators contact your primary care provider?

If the participant answer "YES" to the following question:Have you been hospitalized for psychiatric problem in past year?

If the participant is planning on moving out of the area in the next 36 months

If currently participates in the Band Together exercise program

Positive Callahan cognition screener: If participant fails 2 questions, research coordinator will explain study in detail and ask read-back questions. The participant will be excluded if failed read-back.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1139 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Sciamanna, MD, MPH, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Enhanced Usual Care Plus Exercise Coaching Intervention: Participants will receive the 3 printed pamphlets on fall risks and exercising in groups (same as the controls) plus: (1) an exercise program that includes strength, balance, and aerobic exercises; (2) an exercise coach that provides in-person and telephone support/feedbacks to enhance participation in the exercise program; and (3) regular progress reports sent by coaches by fax/Electronic Health Records every 4 months, to communicate the patient's progress.
  Enhanced Usual Care plus Exercise Coaching: For month 1 of the exercise intervention the investigators will conduct only strength and a few balance exercises to rehabilitate the participants. After the first month, and once the participants feel comfortable, the investigators will incorporate aerobic and additional balance exercises. The investigators will personalize participant programs based on baseline levels and increase them gradually. The exercise session will be conducted 50 minutes 3 times a week. Between sets there is a 60-second break.
  Every month the coach will record steps from the pedometer and record patient adherence to exercise sessions, and every 2 months the coach will measure strength and will track resistance band color from the exercise trackers.
  For the individuals exercising at home, the investigators will distribute the exercise DVDs every 9 months and the coach will continue to contact them, just as if they were joining the group. Coaches will encourage group participation.
Period: Overall Study
Arm/Group | Enhanced Usual Care - Control Group | Enhanced Usual Care Plus Exercise Coaching Intervention
Started | 569 | 570
Completed | 559 | 549
Not Completed | 10 | 21
Not completed — Withdrawal by Subject | 6 | 11
Not completed — Death | 3 | 4
Not completed — Lost to Follow-up | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enhanced Usual Care - Control Group | Enhanced Usual Care Plus Exercise Coaching Intervention | Total
Number analyzed (Participants) | 569 | 570 | 1139
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.2 (6.6) | 73.2 (6.3) | 73.2 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 479 | 482 | 961
  Male | 90 | 88 | 178
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 517 | 508 | 1025
  Black or African-American | 28 | 41 | 69
  Asian | 6 | 3 | 9
  More than One Race | 4 | 8 | 12
  Missing | 14 | 10 | 24
Region of Enrollment [Number; unit: participants]
  United States | 569 | 570 | 1139
Education Level [Count of Participants; unit: Participants]
  Less than high school | 112 | 92 | 204
  College, 1-3 years | 155 | 146 | 301
  College, 4 or more years | 291 | 323 | 614
  Missing | 11 | 9 | 20
Marital Status [Count of Participants; unit: Participants]
  Married/Living with partner | 295 | 299 | 594
  Divorced/Separated | 104 | 86 | 190
  Widowed | 122 | 117 | 239
  Never married | 34 | 55 | 89
  Missing | 14 | 13 | 27
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: Data are missing for 29 participants, 13 in the exercise group and 16 in the control group.
  kg/m^2
    number analyzed (Participants) | 553 | 557 | 1110
    (all) | 28.6 (6.5) | 28.6 (6.5) | 28.6 (6.5)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 129.7 (17.7) | 129.4 (17.8) | 129.5 (17.8)
History of Osteoporosis [Count of Participants; unit: Participants]
  Yes | 261 | 270 | 531
  No | 295 | 292 | 587
  Missing | 13 | 8 | 21
Any fall in past year [Count of Participants; unit: Participants]
  Yes | 271 | 290 | 561
  No | 283 | 262 | 545
  Missing | 15 | 18 | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Fragility Fractures and Serious Fall-Related Injuries (FF/SFI)
Description: Every 4 months the investigators will call the participants asking questions about the main outcome, FF/SFI. A fall calendar will be given to the participant to record all fall events (e.g., date, location). This will help participants to recall falls during the 4 month period. In addition, this will allow medical records to be requested, using a signed authorization form (part of the consent form). The investigators will review all relevant Electronic Health Records (EHR) information, such as hospital and emergency department discharge summaries, outpatient visit notes, consultation notes, physical exam notes, dictated radiologist notes and plain film radiography.
Time Frame: 36 months
Population: All randomized participants
Measure: Number; unit: Participants
Arm/Group | Enhanced Usual Care - Control Group | Enhanced Usual Care Plus Exercise Coaching Intervention
Number analyzed (Participants) | 569 | 570
Participants | 186 | 166
Statistical Analysis 1: Comparison: Enhanced Usual Care - Control Group vs Enhanced Usual Care Plus Exercise Coaching Intervention; Test type: Superiority; p = 0.43, Regression, Cox; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.74 to 1.14] — Enhanced Usual Care - control group vs. Enhanced Usual Care plus Exercise Coaching Intervention

2. Secondary Outcome: Number of Falls and Falls-related Injuries Using the Behavioral Risk Factor Surveillance System (BRFSS)
Description: The investigators will examine the number of falls, and fall-related injuries using two questions from the BRFSS.
Time Frame: 36 months
Measure: Mean (95% Confidence Interval); unit: falls
Arm/Group | Enhanced Usual Care - Control Group | Enhanced Usual Care Plus Exercise Coaching Intervention
Number analyzed (Participants) | 531 | 495
falls | 0.87 [0.79 to 0.95] | 0.84 [0.76 to 0.93]
Statistical Analysis 1: Comparison: Enhanced Usual Care - Control Group vs Enhanced Usual Care Plus Exercise Coaching Intervention; Test type: Superiority; p = 0.50, Regression, Negative Binomial; Incidence Rate Ratio = 1.06, 95% CI 2-sided [0.89 to 1.28] — Enhanced Usual Care - control group vs. Enhanced Usual Care plus Exercise Coaching Intervention

3. Secondary Outcome: Percentage of Participants With Excellent/Very Good Health Using the Patient Reported Outcomes Measurement Information System (PROMIS)
Description: The investigators will use a self-reported health question to assess key patient centered outcomes that the intervention may improve. This question is from the NIH-supported PROMIS. The outcome is categorized as excellent/very good health vs. good/fair/poor health as reported on the single question.
Time Frame: 36 months
Measure: Number; unit: Percentage of participants
Arm/Group | Enhanced Usual Care - Control Group | Enhanced Usual Care Plus Exercise Coaching Intervention
Number analyzed (Participants) | 539 | 506
Percentage of participants | 52.2 | 54.3
Statistical Analysis 1: Comparison: Enhanced Usual Care - Control Group vs Enhanced Usual Care Plus Exercise Coaching Intervention; Test type: Superiority; p = 0.30, Regression, Logistic; Odds Ratio (OR) = 0.89, 95% CI 2-sided [0.72 to 1.11]

4. Secondary Outcome: Assessment of Fear of Falling Using the Falls Efficacy Scale International (FES-I)
Description: The investigators will use the 7-item version of the Falls Efficacy Scale International (FES-I), used to quantify fear of falling in 7 different scenarios. Each item is scored 1-4, with higher scores being associated with greater fear. Total sum score is reported, possible range 7-28.
Time Frame: 36 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Enhanced Usual Care - Control Group | Enhanced Usual Care Plus Exercise Coaching Intervention
Number analyzed (Participants) | 539 | 506
score on a scale | 11.65 [10.96 to 12.33] | 11.11 [10.45 to 11.77]
Statistical Analysis 1: Comparison: Enhanced Usual Care - Control Group vs Enhanced Usual Care Plus Exercise Coaching Intervention; Test type: Superiority; p < 0.01, Mixed Models Analysis; Mean Difference (Final Values) = 0.54, 95% CI 2-sided [0.16 to 0.92] — Enhanced Usual Care - control group vs. Enhanced Usual Care plus Exercise Coaching Intervention

5. Secondary Outcome: Percentage of Participants Meeting Physical Activity Guidelines Using the National Health Interview Survey (NHIS)
Description: The investigators will use 6 questions from the NHIS at baseline and the 36 month follow-up to measure participants' activity level. Percentage of participants with a sum of moderate and vigorous minutes >=150 is reported.
Time Frame: 36 months
Measure: Number; unit: Percentage of participants
Arm/Group | Enhanced Usual Care - Control Group | Enhanced Usual Care Plus Exercise Coaching Intervention
Number analyzed (Participants) | 529 | 487
Percentage of participants | 50.7 | 50.9
Statistical Analysis 1: Comparison: Enhanced Usual Care - Control Group vs Enhanced Usual Care Plus Exercise Coaching Intervention; Test type: Superiority; p = 0.73, Regression, Logistic; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.85 to 1.27] — Enhanced Usual Care - control group vs. Enhanced Usual Care plus Exercise Coaching Intervention

6. Secondary Outcome: Assessment of Physical Function Using PROMIS
Description: The investigators will use 4 physical function questions to assess physical function subscale of PROMIS. Each item ranges 1-5. Total sum score is reported; higher scores are associated with lower levels of physical function. Total sum score range, 4-20.
Time Frame: 36 months
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Enhanced Usual Care - Control Group | Enhanced Usual Care Plus Exercise Coaching Intervention
Number analyzed (Participants) | 539 | 506
Score on a scale | 9.00 [8.28 to 9.72] | 8.77 [8.08 to 9.47]
Statistical Analysis 1: Comparison: Enhanced Usual Care - Control Group vs Enhanced Usual Care Plus Exercise Coaching Intervention; Test type: Superiority; p = 0.27, Mixed Models Analysis; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [-0.18 to 0.62] — Enhanced Usual Care - control group vs. Enhanced Usual Care plus Exercise Coaching Intervention

7. Secondary Outcome: Assessment of Depression Using PROMIS
Description: The investigators will use 4 depression questions to assess key patient centered outcomes that the intervention may improve. These questions are from the NIH-supported PROMIS.
Time Frame: 36 months
Measure: Mean (95% Confidence Interval); unit: score on a scale of 4-20, higher=worse
Arm/Group | Enhanced Usual Care - Control Group | Enhanced Usual Care Plus Exercise Coaching Intervention
Number analyzed (Participants) | 539 | 506
score on a scale of 4-20, higher=worse | 5.62 [5.21 to 6.03] | 5.52 [5.12 to 5.91]
Statistical Analysis 1: Comparison: Enhanced Usual Care - Control Group vs Enhanced Usual Care Plus Exercise Coaching Intervention; Test type: Superiority; p = 0.37, Mixed Models Analysis; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.13 to 0.34] — Enhanced Usual Care - control group vs. Enhanced Usual Care plus Exercise Coaching Intervention

8. Secondary Outcome: Assessment of Anxiety Using PROMIS
Description: The investigators will use 4 anxiety questions to assess key patient centered outcomes that the intervention may improve. These questions are from the NIH-supported PROMIS.
Time Frame: 36 months
Measure: Mean (95% Confidence Interval); unit: score on a scale of 4-20, higher=worse
Arm/Group | Enhanced Usual Care - Control Group | Enhanced Usual Care Plus Exercise Coaching Intervention
Number analyzed (Participants) | 539 | 506
score on a scale of 4-20, higher=worse | 6.21 [5.79 to 6.64] | 6.07 [5.66 to 6.48]
Statistical Analysis 1: Comparison: Enhanced Usual Care - Control Group vs Enhanced Usual Care Plus Exercise Coaching Intervention; Test type: Superiority; p = 0.26, Mixed Models Analysis; Mean Difference (Final Values) = 0.14, 95% CI 2-sided [-0.10 to 0.38] — Enhanced Usual Care - control group vs. Enhanced Usual Care plus Exercise Coaching Intervention

9. Secondary Outcome: Assessment of Loneliness Using PROMIS
Description: The investigators will use 3 loneliness questions to assess key patient centered outcomes that the intervention may improve. These questions are from the NIH-supported PROMIS.
Time Frame: 36 months
Measure: Mean (95% Confidence Interval); unit: score on a scale of 3-9, higher=worse
Arm/Group | Enhanced Usual Care - Control Group | Enhanced Usual Care Plus Exercise Coaching Intervention
Number analyzed (Participants) | 539 | 506
score on a scale of 3-9, higher=worse | 4.19 [3.92 to 4.46] | 4.12 [3.86 to 4.38]
Statistical Analysis 1: Comparison: Enhanced Usual Care - Control Group vs Enhanced Usual Care Plus Exercise Coaching Intervention; Test type: Superiority; p = 0.39, Mixed Models Analysis; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.09 to 0.22] — Enhanced Usual Care - control group vs. Enhanced Usual Care plus Exercise Coaching Intervention

ADVERSE EVENTS:
Time Frame: Data were collected every 4 months for the full 36-month duration of study participation.
Description: Data were collected via structured phone interview which included the use of a calendar used to track falls, specifically.
Arm/Group | Enhanced Usual Care - Control Group | Enhanced Usual Care Plus Exercise Coaching Intervention
All-Cause Mortality (participants affected / at risk) | 22/569 | 30/570
Serious Adverse Events (participants affected / at risk) | 162/569 | 79/570
Other Adverse Events (participants affected / at risk) | 0/569 | 0/570
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enhanced Usual Care - Control Group (N=569) | Enhanced Usual Care Plus Exercise Coaching Intervention (N=570)
Fracture (Musculoskeletal and connective tissue disorders) | 25 (27) | 2 (2)
Elective Joint Replacement (Musculoskeletal and connective tissue disorders) | 18 (18) | 3 (3)
Other Surgery (Surgical and medical procedures) | 14 (16) | 4 (4)
Infection (Infections and infestations) | 20 (23) | 12 (13)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Atrial Fibrillation/Flutter (Cardiac disorders) | 1 (1) | 4 (4)
Heart Failure (Cardiac disorders) | 7 (7) | 3 (4)
Acute Coronary Syndrome / Myocardial Infarction (Cardiac disorders) | 5 (5) | 2 (3)
Stroke / Transient Ischemic Attack / Intracranial Hemorrhage (Cardiac disorders) | 11 (12) | 1 (1)
Fluid / Electrolyte Abnormality (General disorders) | 2 (2) | 3 (3)
Dehydration (General disorders) | 2 (2) | 0 (0)
Imbalance (syncope, dizziness, vertigo) (General disorders) | 3 (3) | 6 (6)
Other (General disorders) | 51 (65) | 37 (45)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-04): https://cdn.clinicaltrials.gov/large-docs/57/NCT02714257/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/57/NCT02714257/ICF_001.pdf